CLINICAL TRIAL: NCT02246803
Title: The Assessment of Progression of Paroxysmal Atrial Fibrillation in Patients After Coronary Artery Bypass Grafting Through Continuous Subcutaneous Monitoring
Brief Title: The Assessment of Progression of Paroxysmal AF After CABG
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Principal Investigator, Alexander Romanov, Meshalkin Research Institute of Pathology of Circulation, Meshalkin Research Institute of Pathology of Circulation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AF-Progress
Record Dates: First submitted 2014-09-19; First posted 2014-09-23 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Paroxysmal Atrial Fibrillation, Coronary Artery Disease
Keywords: paroxysmal atrial fibrillation, CABG, pulmonary vein isolation
MeSH Terms: conditions — Atrial Fibrillation; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CABG+pulmonary vein isolation (Active Comparator): CABG+pulmonary vein isolation procedure
  Interventions: Procedure: CABG+Pulmonary vein isolation procedure
- Isolated CABG (Active Comparator): Isolated CABG procedure
  Interventions: Procedure: Isolated CABG

INTERVENTIONS:
Procedure: CABG+Pulmonary vein isolation procedure — Coronary artery bypass (CABG) using cardio-pulmonary bypass (CBP) and occlusion. Concomitant pulmonary vein isolation in CBP prior to occlusion and CABG
  Arms: CABG+pulmonary vein isolation
Procedure: Isolated CABG — Coronary artery bypass (CABG) using cardio-pulmonary bypass (CBP) and occlusion.
  Arms: Isolated CABG

SUMMARY:
The aim of this study is a comparative evaluation of progression of paroxysmal atrial fibrillation in patients with coronary artery disease after isolated CABG and CABG combined with pulmonary vein isolation.

Hypothesis of the study - patients with paroxysmal atrial fibrillation and coronary artery disease after CABG in combination with isolation of the pulmonary veins have a better outcomes for the progression of AF compared with patients undergoing isolated CABG.

DETAILED DESCRIPTION:
This is a single blinded prospective randomized study involving 72 patients with paroxysmal AF and coronary artery disease. 72 patients are required to have a 80% chance of detecting, as significant at the 5% level, an increase in the primary outcome measure by 10% in the CABG + pulmonary veins isolation group over isolated CABG group. Patients are divided into two groups, group I - isolated CABG (36 patients), and group II - CABG and pulmonary veins isolation (36 patients). Randomization is conducted by using accidental sampling before operation. The blinding process is applied to a patient, who is informed about received coronary artery bypass grafting, but don't know about pulmonary vein isolation. Subcutaneous cardiac monitor is implanted to all patients for cardiac rhythm monitoring.

ELIGIBILITY:
Inclusion Criteria:

* American College of Cardiology (ACC)/ American Heart Association (AHA) -Indications for CABG
* At least 2 ECG-verified (12-channel ECG, Holter telemetry) symptomatic paroxysmal atrial fibrillation episodes within last 12 months
* The patient's consent to participate in the study

Exclusion Criteria:

* Intolerance of antiarrhythmic drugs
* Heart valve disease requiring invasive treatment
* Left atria more than 6.5 cm
* Prior cardiac surgery
* Active pacemaker treatment
* Active anti-arrhythmic treatment (AAD) class I and III
* Contraindication to oral anticoagulant/heparin treatment
* Ejection fraction less than 30 % (EF < 30 %) assessed by transthoracic echocardiography

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Progression of atrial fibrillation | up to 36 months
  Combined indicator consist of recurrence of AF, increased frequency of AF, progression to persistent AF.
  Atrial fibrillation is defined as atrial fibrillation paroxysm lasting at least 60 seconds. Patients with AF>0.5% were classified as non-responders.

SECONDARY OUTCOMES:
Hospitalization due to atrial fibrillation after surgery | Within three years after surgery
  All cases of hospitalization due to atrial fibrillation after surgery
Cardiovascular events | Within three years after surgery
  All cases of stroke, cardiac infarction, thromboembolism, bleeding and death

CONTACTS AND LOCATIONS:
Locations (1):
- Meshalkin State Research Institute of Circulation Pathology, Novosibirsk, Russia